CLINICAL TRIAL: NCT05525871
Title: Experimental Study to Evaluate the Effects of Effects of a Sports Supplement Based on Nitrates and Citrulline Malate on Performance in Professional Soccer Players
Brief Title: Effects of Nitrates and Citrulline Malate on Performance in Professional Professional Soccer
Acronym: NiCiFut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00027
Record Dates: First submitted 2022-08-09; First posted 2022-09-02 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2022-07

CONDITIONS: Supplementation
Keywords: Nitrates; Citrulline malate; Soccer
MeSH Terms: interventions — Nitrates; citrulline malate; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrates and Citrulline Malate (Experimental): Gel elaborated from fruit puree with high polyphenol content, with the addition of nitrates and citrulline malate as study supplements. addition of nitrates and citrulline malate as study supplements.
  Interventions: Dietary Supplement: Nitrates and Citrulline Malate
- Control product (Placebo Comparator): Consumption of placebo product (Fruit puree)
  Interventions: Dietary Supplement: Control product

INTERVENTIONS:
Dietary Supplement: Nitrates and Citrulline Malate — Female soccer players should consume the experimental product for 30 days to evaluate the efficacy of a sports supplement high in nitrates combined with citrulline malate in the improvement of performance in high-intensity intermittent exercise.
  high intensity
  Arms: Nitrates and Citrulline Malate
Dietary Supplement: Control product — Fruit puree
  Arms: Control product

SUMMARY:
Randomized, single-center, parallel, team-stratified, stratified experimental study to evaluate the efficacy of a high sports supplement in improving high-intensity intermittent exercise performance in professional female soccer players.

DETAILED DESCRIPTION:
Subjects who meet the selection criteria will be randomly assigned to each of the study groups (investigational product or placebo, depending on the group to which they have been assigned).

The product to be consumed will be Nitrates and Citrulline Malate. Participants will consume the product for 30 days. The intake should be done two hours before each training session and the same dose will be consumed.

The women's soccer players will perform a stress test with gas analysis to measure performance, as well as a Wingate test without consumption of the products. Five days later, the players will perform the Yo-Yo IR1 test in the field and will repeat the same tests performed at the beginning of the test after product consumption.

ELIGIBILITY:
Inclusion Criteria:

* Present at the time of signing the informed consent at the age between 18 and 40 years.
* Female.
* Healthy subjects without any chronic disease.
* Volunteers capable of understanding the clinical study, willing to give their written informed. consent and comply with the procedures and requirements of the study. and requirements of the study.

Exclusion Criteria:

* Players who change teams during the experimental study.
* Smoking subjects.
* Subjects using mouthwashes during the study.
* Subjects with a history of drug, alcohol or other substance abuse or other factors that limit their ability to cooperate during the study. factors that limit their ability to cooperate during the study.
* Subjects whose status makes them ineligible for the study, at the discretion of the investigator discretion of the investigator.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Aerobic and anaerobic thresholds - VO2max | Change in initial maximal oxygen consumption at 30 days
  Measured with a gas analyzer
Fatigue in jumping | Change in initial jump fatigue at 30 days
  Measured with a contact platform
Anaerobic capacity | Change in baseline anaerobic capacity at 30 days
  Measured with a Monark cycloergometer

SECONDARY OUTCOMES:
Microcapillary blood | It will be measured on two different occasions. Day one and 30 days later.
  This test provides biochemical variables (ABL90FLEX) with 70 ml of capillary blood.
Lactate | It will be measured on two different occasions. One on the first day (without intake of product ) and 30 days later, the same measurements but after having consumed the product
  Lactate levels will be measured using the Lactate Pro
Safety variables | It will be measured on two different occasions. Day one and 30 days later.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain